CLINICAL TRIAL: NCT06715995
Title: Effects of Endogenous Gamma Light Stimulation on Brain Oscillations in Cognitively-normal Older Adults: a Randomized, Placebo-controlled, Double-blind Study
Brief Title: Effects of Endogenous Gamma Light Stimulation on Brain Oscillations in Cognitively-normal Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Aleddra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202401421B0A3
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: EEG Brain Oscillations; Alzheimer's Disease (AD); Cognitively Normal Older Adults
Keywords: Endogenous gamma; EEG rhythms; Resting-state EEG (rs-EEG); Alzheimer's disease (AD); Cognitive function; non-flickering light

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- endogenous gamma light (Active Comparator): This device is an LED light source table lamp with a vertical surface measuring 16 cm by 22 cm. It will be positioned within arm's reach, approximately 50 cm from the participant, to ensure continuous exposure to the light stimulation. The active device delivers endogenous gamma light stimulation.
  Interventions: Device: Gamma Wave Stimulation Table Lamp (Aleddra, Inc., USA)
- Sham (70Hz) gamma light (Sham Comparator): The sham device is identical in appearance to the active device. It will be positioned within arm's reach, approximately 50 cm from the participant, to ensure continuous exposure to the light stimulation. The sham device delivers 70 Hz light stimulation.
  Interventions: Device: Gamma Wave Stimulation Table Lamp (Aleddra, Inc., USA)

INTERVENTIONS:
Device: Gamma Wave Stimulation Table Lamp (Aleddra, Inc., USA) — Participants will receive light stimulation using the Gamma Wave Stimulation Table Lamp (Aleddra, Inc., USA) for 1 hour per day, 7 days a week, over 4 weeks, for a total of 28 hours.

SUMMARY:
This study aims to evaluate the effects of endogenous gamma non-flickering light stimulation on resting-state EEG rhythms and cognitive function in cognitively healthy older adults. Specifically, it will assess the immediate and long-term effects of this stimulation on brainwave activity and cognitive performance. The study will explore the potential of gamma light stimulation as a non-pharmacological intervention for cognitive decline in aging populations.

DETAILED DESCRIPTION:
Some Alzheimer's disease (AD) studies have investigated the effects of gamma-frequency light stimulation on healthy older adults and AD patients; they have several limitations, including small sample sizes, short intervention durations, the use of flickering light (which may cause discomfort), and lack of rigorous randomized controlled trials. The aim of this study is to address these gaps by conducting a randomized, placebo-controlled, double-blind trial.

This study will recruit 52 cognitively healthy older adults aged 55 and above (N= 52). Participants will be randomly assigned to either the experimental group (N=26), receiving endogenous gamma non-flickering light stimulation, or the control sham group (N=26), receiving 70 Hz non-flickering light stimulation. The intervention will consist of 1 hour of daily stimulation, 7 days a week, for a total of 4 weeks (28 hours). Both participants and outcomes assessors will remain blinded to group allocation.

Resting-state EEG and cognitive assessments will be conducted at three time points: prior to the intervention (T1), post one-hour intervention (T2), and post one-month intervention (T3). Resting-state brainwave activity will be the primary outcome, with data collected at all three time points (T1, T2, and T3). As secondary outcomes, cognitive assessments will be administered at T1 and T3. Adverse events will also be recorded by participants immediately following each light stimulation session.

The primary aim of this study is to assess the immediate (T2 relative to T1) and long-term (T3 relative to T1) effects of endogenous gamma light stimulation on resting-state brainwave activity. Secondary objectives include evaluating cognitive performance and assessing the safety, user acceptance, and adherence to the intervention device. The results of this study will provide valuable insights into the potential of endogenous gamma light stimulation as a non-pharmacological intervention for cognitive decline in aging populations.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age over 55 years old.
* 2. The Cognitive Abilities Screening Instrument (CASI) score is within normal ranges adjusted for age and education.
* 3. Participants have no history of severe neurological or psychiatric disorders (such as stroke, epilepsy, depression, migraine, etc.) that could affect cognitive function.
* 4. Participants have not used drugs that may affect cognitive function (e.g., benzodiazepines, anticholinergic medications, etc.).
* 5. Participants with normal or corrected vision (e.g., glasses or contact lenses) to normal levels.
* 6. Voluntary to sign the Informed Consent Form.

Exclusion Criteria:

* 1. Participants enrolled in any cognitive enhancement study within the past two months.
* 2. Participants with a history of disease that could affect cognitive function (e.g., cancer, autoimmune diseases, etc.).
* 3. Pregnant, or planning to become pregnant.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gamma brain oscillations. | baseline (T1), post one-hour intervention (T2), post one-month intervention (T3)
  Gamma (31-100Hz) brain oscillations obtained through resting-state EEG will evaluate the changes of gamma light stimulation intervention.

SECONDARY OUTCOMES:
Change score of the Cognitive Abilities Screening Instrument (CASI). | baseline (T1), post one-month intervention (T3)
  CASI will be applied to measure the participant's general cognitive ability. The range of score is 0 to 100, with a higher score indicating better performance.
Change score of the Chinese version Verbal Learning Test (CVVLT). | baseline (T1), post one-month intervention (T3)
  A nine-item of CVVLT (total recall, delayed recall) will be applied to measure the participant's memory ability, with a higher score indicating better performance.
Change score of the WMS-III logical memory test | baseline (T1), post one-month intervention (T3)
  WMS-III logical memory test (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 25 for each recall trial, with a higher score indicating better performance
Change score of the Taylor Complex Figure Test (TCFT). | baseline (T1), post one-month intervention (T3)
  TCFT (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 36 for each recall trial, with a higher score indicating better performance.
Performance changes of the Trail Making Test Form A/B (TMT-A/B). | baseline (T1), post one-month intervention (T3)
  TMT-A/B will be applied to measure participant's attention and executive function.
  The number of seconds to complete each trial and the number of errors would be recorded, with a higher value indicating greater impairment.
Subjective cognition decline complaint survey. | baseline (T1), post one-month intervention (T3)
  A 14-item Subjective Memory Complaints Questionnaire measured memory impairment. The response was restricted to either "Yes" or "No".
Change score of the category Verbal Fluency Test (VFT). | baseline (T1), post one-month intervention (T3)
  The category VFT will be applied to measure the participant's language and executive function, with a higher score indicates better performance.
Safety/Adverse event outcome measure. | Throughout the one-month intervention
  Adverse events, such as fatigue, headache, dizziness, dazzling, ocular pain, and others, will be recorded using a 6-point Likert scale ranging from 'not at all' to 'extremely uncomfortable' (0 = not at all, 1 = minimal discomfort, 2 = mild discomfort, 3 = tolerable, 4 = severe discomfort, 5 = extreme discomfort).
  Participants will report adverse events (such as fatigue, headache, dizziness, dazzling, ocular pain, and others) using a 6-point Likert scale ranging from 'not at all' to 'extremely uncomfortable' after each light stimulation session.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No